CLINICAL TRIAL: NCT07136857
Title: Study To Assess Response to Eptacog Beta iN Patients With Glanzmann THromboasthenia (STRENGTH )
Brief Title: Eptacog Beta in Glanzmann's (HeT_LFB-Strength-Study_FID531)
Acronym: STRENGTH
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Laboratoire Français du Fractionnement et des Biotechnologies (LFB BIOTECHNOLOGIES) (Unknown)
Responsible Party: Principal Investigator, Karen L. Zimowski, Assistant Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00009481; 2025P010364 (Other: Emory IRB)
Record Dates: First submitted 2025-08-15; First posted 2025-08-22 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Glanzmann Thrombasthenia
Keywords: Severe Bleeding; Prevention of Bleeding; Eptacog beta (EB)
MeSH Terms: conditions — Thrombasthenia; Hemorrhage | interventions — recombinant FVIIa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Eptacog beta (Experimental): For the initial 3 months, participants will be in a non-interventional phase and receive standard-of-care on-demand therapy for acute bleeding at their hematologist's discretion. Following this non-interventional phase, they will use eptacog beta on-demand to treat acute bleeding for 6 months. Throughout the study, they will log bleeding events and management in a diary. Hemostatic efficacy after treatment will be assessed using a 4-point hemostasis efficacy scale.
  Participants will have the option to re-consent for an exploratory phase, adding 6 months to their time on the study (total of 15 months). For those entering the optional extension phase, eptacog beta will be routinely administered for bleed prophylaxis. The treating hematologist will determine the best method/location for infusions. The number of bleeding events over time will be compared between the prophylaxis phase and the on-demand phase.
  Interventions: Drug: EPTACOG BETA

INTERVENTIONS:
Drug: EPTACOG BETA — Eptacog beta (SEVENFACT®; EB) is a lyophilized powder in single-use vials (1, 2, or 5 mg) of coagulation factor VIIa (recombinant)-jncw. It is reconstituted with sterile water (provided in the kit) and administered intravenously.
  SEVENFACT® may be administered by a healthcare provider (HCP) at the study site or home, or by a trained participant/caregiver. Participants will be monitored in a healthcare facility for 60 minutes after the first dose for hypersensitivity.
  Other Names: SEVENTFACT®; EB

SUMMARY:
This study is evaluating an investigational drug, eptacog beta (EB), for the treatment and prevention of acute bleeding episodes in people with Glanzmann Thrombasthenia, a rare inherited bleeding disorder. Eptacog beta (EB) is not currently approved by the U.S. Food and Drug Administration (FDA) for this condition.

The study will assess the effectiveness and safety of eptacog beta (EB) when used to treat serious bleeding events, and in an optional phase, when used routinely to prevent bleeding. During the first three (3) months, participants will manage any bleeding episodes with their standard treatment (e.g., factor products or platelet transfusions). After this initial period, they will use the study drug to treat serious bleeding events.

Participants will have approximately 4 to 5 visits with their hematologist over the 9-month study period. They will also be asked to complete a diary documenting bleeding episodes and treatments, and to answer questions about how bleeding affects their daily life. Blood samples will be collected to monitor their condition and any potential side effects of the study drug.

At the end of the main study, participants will have the option to enter an optional extension phase, where they will receive routine intravenous infusions of the study drug 2 to 3 times per week for 6 months to help prevent future bleeding episodes and complications.

DETAILED DESCRIPTION:
This study aims to investigate eptacog beta (EB), a new form of recombinant activated factor VIIa, for bleeding management in persons with Glanzmann thrombasthenia regardless of platelet refractoriness status.

Investigators will enroll six (6) people (adult or pediatric) with Glanzmann thrombasthenia (GT) who have a severe bleeding phenotype (defined as ≥ 2 treated bleeding events in the past 12 months, ≥ 1 hospitalization for bleeding or severe anemia or requiring prophylactic therapy to prevent bleeding). Initially, a retrospective chart review will collect data regarding bleeding events and their management over the previous 6 months before enrollment.

The initial 3 months of this trial will be a non-interventional phase during which time, participants will receive standard-of-care on-demand therapy for acute bleeding events at the discretion of their hematologist. They will complete a diary logging their bleeding events and their management. Hemostatic efficacy following acute bleed treatment will be evaluated using a 4-point hemostasis efficacy score.

Following this initial non-interventional phase, participants will use eptacog beta (EB) 75 mcg/kg/dose every 3 Hours for the management of breakthrough bleeding episodes that are not responsive to local hemostatic control and anti-fibrinolytic therapies, with the precise frequency of infusions and duration of treatment at the discretion of the subject's treating physician. This on-demand interventional phase will last 6 months. During this time, participants will log their acute bleeding episodes and management. At varying time points following a dose of EB, participants will complete a 4-point hemostasis scale assessing the efficacy of EB in controlling bleeding.

Following the 6-month interventional on-demand phase, participants may choose to continue in an interventional prophylaxis arm.

ELIGIBILITY:
Inclusion Criteria:

* Adult or Pediatric persons with inherited Glanzmann thrombasthenia (see diagnostic criteria below)
* Severe bleeding phenotype
* Adequate hepatic function
* Adequate renal function
* Adults subject (≥18 years of age) or caregiver (parent or legally authorized representative) for minor subjects, subjects with cognitive impairment, or subjects with impaired decision-making capacity have provided written informed consent, and the participant has given consent/assent (if applicable)
* Ability to speak, read, and understand the English language

Exclusion Criteria:

* Thrombocytopenia (platelet count < 100k)
* Acquired Glanzmann thrombasthenia secondary to autoimmune disease, malignancy, or medication
* Inherited or acquired bleeding diathesis other than Glanzmann thrombasthenia
* Have a history of venous or arterial thrombotic event within 2 years of study enrollment
* Active malignancy
* Known or suspected hypersensitivity to rabbits, rabbit protein, other forms of rFVIIa, or to any of the EB excipients
* Have received an investigational drug within 30 days or within 5 half-lives of that investigational drug (whichever is longer) or are expected to receive such a drug during participation in this study
* Be using aspirin, non-steroidal anti-inflammatory drugs (NSAIDS), herbs, natural medications, or other drugs with platelet inhibitor properties for the duration of the study
* Be using or administered anticoagulant agents for the duration of the study
* Have any life-threatening disease or other disease or condition which, according to the investigator's judgement, could imply a potential hazard to the patient, or interfere with the study participation or study outcome
* Use of systemic immunomodulators at enrollment or planned use during the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2025-10-02 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of bleeding events successfully treated within 24 hours of the first Eptacog Beta (EB) administration | 24 hours after the first EB dose administration
  Proportion of acute bleeding events successfully treated with EB within 24 hours of the first EB administration based on an "excellent or good" response on a 4-point hemostatic efficacy scale and without rebleeding before 36 hours.
  Hemostatic Efficacy Scale:
  None = No effect; bleeding unchanged or worsened; continued treatment needed.
  Moderate = Some effect (e.g., pain decreased, bleeding signs improved) but bleeding continued; further treatment needed.
  Good = Bleeding symptoms are largely reduced but not completely resolved; no further EB infusions are needed.
  Excellent = Full relief of bleeding symptoms; no additional EB infusion required.
Number of bleeding events over the study period | 6 months following the start of the interventional prophylaxis phase
  The number of bleeding events occurring while receiving routine EB prophylaxis will be compared with the number of bleeding events that occurred during on-demand therapy.
  *This outcome applies only to the optional interventional prophylaxis phase.

SECONDARY OUTCOMES:
Number of treatment-Emergent Adverse Events and Clinically Significant Laboratory Abnormalities | 6 months following the start of EB administration for each study phase
  Safety of EB will be measured by the number of treatment-emergent adverse events, treatment-emergent serious adverse events, and treatment-emergent potentially clinically significant laboratory values reported during the interventional phases compared to those reported during the non-interventional observational phase.
EuroQol five-dimensional questionnaire for youth (EQ-5D-Y) score for participants 4-15 years of age. | Baseline, 9 and 15 months after baseline
  The EQ-5D-Y-5L is a child-friendly, five-dimension, five-level instrument assessing: Mobility, Looking After Myself, Doing Usual Activities, Having Pain or Discomfort, and Feeling Worried, Sad, or Unhappy.
  Each dimension has five response levels (1 = no problems to 5 = extreme problems/unable to do). Respondents select one statement per dimension describing their health on the assessment day, forming a 5-digit profile summarizing their health state. For example, code 11234 indicates no problems with mobility or looking after myself, slight problems doing usual activities, some pain or discomfort, and feeling very worried, sad, or unhappy. Higher scores reflect greater severity.
  *15 months applies to the optional phase only.
EuroQol five-dimensional 5 Level (EQ-5D-5L) score for participants ≥16 years | Baseline, 9 and 15 months after baseline
  The EuroQol 5 Dimension 5 Level (EQ-5D-5L) is a self-report survey that measures quality of life across 5 domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. It captures how people feel across five dimensions, each of which has five levels: 1 = no problems to 5 = extreme problems/unable to do. The five answers produce a unique 5-digit health state, for example, 11234, that describes the young person's health state. For example, the code 11234 describes a health state where there are no problems with walking about (mobility) or looking after myself, a little bit of a problem with doing usual activities, some pain or discomfort, and feeling really worried, sad, or unhappy.
  *15 months applies to the optional phase only.
Patient Reported Outcomes Measurement Information System (PROMIS) fatigue short form for adults | Baseline, 9 and 15 months after baseline
  The PROMIS Fatigue item banks assess a range of self-reported symptoms, from mild subjective feelings of tiredness to an overwhelming, debilitating, and sustained sense of exhaustion that likely decreases one's ability to execute daily activities and function normally in family or social roles. Fatigue is divided into the experience of fatigue (frequency, duration, and intensity) and the impact of fatigue on physical, mental, and social activities. The fatigue short forms are universal and assess fatigue over the past seven days. PROMIS measures use a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population. On the T-score metric:
  A score of 40 is one SD lower than the mean of the reference population. A score of 60 is one SD higher than the mean of the reference population. Higher scores equal more fatigue.
  *15 months applies to the optional phase only.
PROMIS fatigue short form (pediatric version) | Baseline, 9 and 15 months after baseline
  The PROMIS Pediatric Fatigue Short Form will be used to assess fatigue based on age: self-report (ages 8-17) and parent-proxy (ages 5-17). It measures fatigue symptoms and their impact on physical, mental, and social activities over the past 7 days. Items reflect both the frequency and severity of fatigue. Scores are reported as T-scores (mean = 50, SD = 10) based on a reference population. A higher T-score indicates greater fatigue (e.g., 60 = 1 SD above the mean). This measure captures the participant's ability to carry out daily activities and participate in usual roles.
  *15 months applies to the optional phase only.
Menstrual impact questionnaire (MIQ) score | Baseline, 9 and 15 months after baseline
  The MIQ was developed to assess the effect of heavy menstrual bleeding (menorrhagia) on various aspects of a woman's quality of life (QoL). It is a brief, 6-item patient-reported outcome measure that focuses on: Perceived amount of blood loss, limitations in work, physical and social activities, and changes due to treatment. Each item is rated on a 6-point scale, indicating the severity of impact (e.g., 0 = no effect, up to 5 = severe effect).
  Total Score = Sum of all 6 items (range 0-30), with higher scores reflecting a greater negative impact of menorrhagia on daily life.
Exogenous thrombin potential (ETP) following ex vivo EB | Baseline (pre-infusion)
  ETP concentration following ex vivo spiking in various concentrations of EB. Samples will be compared to baseline participants and healthy control samples.
Lag time and time to peak thrombin following ex vivo EB | Baseline (pre-infusion)
  Lag time and time to peak thrombin following ex vivo spiking in various concentrations of EB. Samples will be compared to baseline participants and healthy control samples.
Peak thrombin levels following ex vivo EB | Baseline (pre-infusion)
  Peak thrombin levels following ex vivo spiking in various concentrations of EB. Samples will be compared to baseline participants and healthy control samples.
ETP levels following in vivo EB | Preinfusion, 30 and 60 minutes following the first EB infusion
  ETP thrombin levels at 30 and 60 minutes following in vivo infusion of EB. Samples will be compared to pre-infusion baseline participant and healthy control samples.
Lag time and time to peak thrombin following in vivo EB infusion | Preinfusion, 30 and 60 minutes following the first EB infusion
  Lag time and time to peak thrombin at 30 and 60 minutes following in vivo infusion of EB. Samples will be compared to pre-infusion baseline patient PRP and healthy control samples.
Peak thrombin following in vivo EB infusion | Preinfusion, 30 and 60 minutes following the first EB infusion
  Peak thrombin at 30 and 60 minutes following in vivo infusion of EB. Samples will be compared to pre-infusion baseline patient platelet-rich plasma (PRP) and healthy control samples.
Clotting time (CT) and clotting formation time (CFT) following in vivo EB infusion | Preinfusion, 30 and 60 minutes following the first EB infusion
  CT and CFT will be measured using rotational thromboelastometry following ex vivo spiking with various concentrations of EB. Samples will be compared to baseline samples and healthy control samples.
Maximum clot firmness (MCF) following in vivo EB infusion | Preinfusion, 30 and 60 minutes following the first EB infusion
  MCF will be measured using rotational thromboelastometry following ex vivo spiking with various concentrations of EB. Samples will be compared to baseline samples and healthy control samples.
Alpha angle following ex vivo EB | Preinfusion, 30 and 60 minutes following the first EB infusion
  The alpha angle will be measured using rotational thromboelastometry following ex vivo spiking with various concentrations of EB. Samples will be compared to baseline samples and healthy control samples.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Zimowski, MD, Principal Investigator — Emory University
Locations (1):
- Arthur M. Blank Hospital | Children's Healthcare of Atlanta, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No